CLINICAL TRIAL: NCT07198906
Title: A NEW WAY TO DETECT ACUTE KIDNEY INJURY AFTER CARDIAC SURGERY
Brief Title: A NEW WAY TO DETECT ACUTE KIDNEY INJURY
Acronym: VEX-CARDS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/213/OB; 2023-A02389-36 (Other: ANSM)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Renal Failure
Keywords: heart surgery; postoperative complication
MeSH Terms: conditions — Acute Kidney Injury; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — As part of routine intensive care, blood samples are taken daily to measure creatinine, blood ionogram, NT-pro-BNP, and troponin levels. The results of these measurements will be analyzed as part of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Determination of VEXUS score and onset of chronic renal failure — The aim is to prospectively evaluate the association between the ultrasound score (VEXUS) and the occurrence of acute renal failure post-operatively following cardiac surgery. The VEXUS (Venous Excess UltraSound) score is an ultrasound tool used in medicine to assess systemic venous congestion, i.e. excess pressure in the venous system linked to volume overload or right heart failure. The VEXUS score relies on ultrasound of the inferior vena cava (IVC) to assess the extent of congestion in this vein. score 0 : Normal IVC + Normal Dopplers; score 1 : Dilated IVC + altered hepatic venous Doppler, but normal portal vein; score 2 : Portal vein shows significant pulsatility; score 3 : Severe pulsatility + marked alteration of hepatic and portal flow

SUMMARY:
Acute renal failure after cardiac surgery is a common postoperative complication, affecting approximately 20% of patients. It is associated with an increase in short-term mortality and an increase in hospital stay; but is also associated with an increase in long-term mortality of up to 30% at 5 years, even if renal function recovers upon discharge.

Its origin is multifactorial: intraoperative hypoperfusion, including hemodynamic variations related to extracorporeal circulation or bleeding, postoperative hypoperfusion related to cardiogenic or vasoplegic shock, ischemia-reperfusion phenomena leading to cell lysis or inflammation at the tubular level, inflammation and oxidative stress related to extracorporeal circulation, and hemolysis are the main causes.

Hydro-sodium overload and associated venous congestion is also one of the etiologies of acute renal failure in post-operative cardiac surgery and is associated with increased mortality. The proposed pathophysiological mechanism is based on the decrease in renal tissue perfusion pressure due to the increase in venous pressure. In the extreme, the increase in pressure in the renal capsule could lead to true renal ischemia due to engorgement. This renal congestion can be diagnosed based on clinical signs, biological signs (such as NT-pro-BNP) or by monitoring by central venous pressure (CVP). However, these statistical tools have low diagnostic performance, and new tools based on ultrasound and Doppler are being developed. Indeed, alterations in venous flow in the renal, suprahepatic and portal veins, reflecting the increase in pressures there, are associated with the onset of acute renal failure in post-operative cardiac surgery.

DETAILED DESCRIPTION:
More recently, a retrospective postoperative cardiac surgery study assessed venous congestion using the VEXUS (Venous Excess UltraSound) composite score. This score explores the diameter of the inferior vena cava (IVC) and venous flows in the hepatic, portal, and renal veins, and is associated with acute renal failure. Its diagnostic performance is based on the joint analysis of all Doppler flows and offers better diagnostic performance than isolated CVP measurement.

The primary objective of this study is to prospectively investigate this ultrasound score and its association with the development of acute renal failure postoperatively after cardiac surgery. Due to the morbidity and mortality associated with renal failure described above, a secondary objective of the study is to investigate the association between the VEXUS score and the development of chronic renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing valve surgery and/or bypass surgery under cardiopulmonary bypass (CPB).
* Patient who has read and understood the information letter and does not object to participating in the study.
* Member of or beneficiary of a social security scheme.

Exclusion Criteria:

* Age under 18 years
* Severe chronic kidney disease with glomerular filtration rate (GFR) < 30 mL/min/1.73 m² and/or requiring dialysis treatment
* Kidney, heart, and liver transplant recipients
* Acute kidney failure at the time of inclusion, defined by KDIGO criteria
* Coronary artery bypass grafting without CPB
* Conditions that may interfere with portal and liver Doppler imaging (cirrhosis, suspected cirrhosis, portal thrombosis)
* Mechanical left ventricular support
* Circulatory support such as ECLS
* Pregnant women
* Patient refusal
* Protected incapacitated persons (judicial protection, guardianship, curatorship, deprivation of liberty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient undergoing valve surgery and/or bypass surgery under extracorporeal circulation (ECC).
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
To study the association between the VEXUS score and the occurrence of acute renal failure post-operatively after cardiac surgery. | visit Hour no. 02, i.e. 2 hours after the intervention; visit Day 1 and visit Day 2
  Onset of acute renal failure characterized by a score greater than or equal to KDIGO 1. (KDIGO 1 : Creatinine increased by >26.5 µmol/L or 1.5-1.9 times the reference value, Diuresis <0.5 mL/kg/h for 6-12 hours; KDIGO 2 : Creatinine x 2-2.9 compared to the reference value, Diuresis < 0.5/mL/kg/h for > 12h; KDIGO 3 : Creatinine x 3 or increase of >353.6 µmol/L compared to the reference value Use of extra-renal replacement therapy, Diuresis < 0.3 mL/kg/h for > 24 hours or anuria for > 12 hours.)

SECONDARY OUTCOMES:
Study of the correlation or association between the VEXUS score and - the value of Central Venous Pressure (CVP) | visit Hour no. 02, i.e. 2 hours after the intervention; visit Day 1 and visit Day 2
  Studying the correlation between the VEXUS score and PVC allows us to validate or not the VEXUS as a reliable non-invasive tool for assessing venous congestion.
Study of the correlation or association between the VEXUS score and the NT-pro-BNP level | visit Hour no. 02, i.e. 2 hours after the intervention; visit Day 1 and visit Day 2
  Studying the relationship between VEXUS score and NT-proBNP (biomarker of cardiac volume overload) helps determine whether venous ultrasound can be a reliable substitute for the biomarker to detect volume congestion, especially in critically ill patients.
Study of the correlation or association between the VEXUS score and the Hydro-sodium balance in intensive care | visit Hour no. 02, i.e. 2 hours after the intervention; visit Day 1 and visit Day 2
  to determine whether the VEXUS score, which reflects venous congestion assessed by ultrasound, is correlated or associated with the hydro-sodium balance, i.e. the quantity of liquid and sodium retained or eliminated by a patient in intensive care
Study of the correlation or association between the VEXUS score and The time of the first dose of diuretics administered | visit Hour no. 02, i.e. 2 hours after the intervention; visit Day 1 and visit Day 2
  Determine whether a high VEXUS score is associated with early administration of diuretics, which would allow us to Validate VEXUS as a therapeutic decision-making tool
Study of the correlation or association between the VEXUS score and The onset of chronic renal failure (assessed at 3 months) | visit month 3
  To determine whether the VEXUS score, used from hospitalization, can predict chronic renal evolution at 3 months.
Study of the correlation or association between the VEXUS score and The length of hospitalization | Visit 12 months
  To determine whether the VEXUS score, measured at the beginning or during hospitalization, is correlated or associated with the total length of hospital stay (unity : day)
Study of the correlation or association between the VEXUS score and The onset of chronic renal failure (assessed at 12 months) | visit month 12
  To determine whether the VEXUS score, used from hospitalization, can predict chronic renal evolution at 12 months.
Study of the correlation or association between the VEXUS score and The mortality (assessed at 3 months) | visit month 3
  Validating VEXUS as a prognostic marker with mortality at 3 months.
Study of the correlation or association between the VEXUS score and The mortality (assessed at 12 months) | visit month 12
  Validating VEXUS as a prognostic marker with mortality at 12 months.
Study of the correlation or association between the VEXUS score and The quality of life (assessed at 3 months) | visit month 3
  Validate VEXUS as a prognostic marker of 3-month mortality with EQ-5D-5L quiz. The EQ-5D-5L is a standardized questionnaire designed to measure health-related quality of life (HRQoL). Five levels are assessed: Mobility; Self-care; Usual activities; Pain/discomfort and Five levels are assessed: Anxiety/depression. Each dimension has 5 severity levels, rated from 1 to 5. (level 1 : No problem; level 2 : Mild problem; level 3 : Moderate problem; level 4 : Severe problem; level 5 : Extreme disability / very severe problem). The patient's overall health status is determined on a scale of 0 to 100 (0 = worst imaginable health status; 100 = best imaginable health status)
Study of the correlation or association between the VEXUS score and The quality of life (assessed at 12 months) | visit month 12
  Validate VEXUS as a prognostic marker of 12-month mortality with EQ-5D-5L quiz. The EQ-5D-5L is a standardized questionnaire designed to measure health-related quality of life (HRQoL). Five levels are assessed: Mobility; Self-care; Usual activities; Pain/discomfort and Five levels are assessed: Anxiety/depression. Each dimension has 5 severity levels, rated from 1 to 5. (level 1 : No problem; level 2 : Mild problem; level 3 : Moderate problem; level 4 : Severe problem; level 5 : Extreme disability / very severe problem). The patient's overall health status is determined on a scale of 0 to 100 (0 = worst imaginable health status; 100 = best imaginable health status)

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.